CLINICAL TRIAL: NCT06330324
Title: Reproductive Options in Inherited Skin Diseases: an International Observational Cohort Study
Brief Title: Reproductive Options in Inherited Skin Diseases
Acronym: REPRO-ISD
Status: Enrolling by invitation | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: METC 2023-0182
Record Dates: First submitted 2024-03-11; First posted 2024-03-26 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Ichthyosis; Palmoplantar Keratoses; Epidermolysis Bullosa; Ectodermal Dysplasia; Basal Cell Nevus Syndrome; Birt-Hogg-Dube Syndrome; Tuberous Sclerosis; Xeroderma Pigmentosum; Cutis Laxa; Albinism
MeSH Terms: conditions — Ichthyosis; Keratoderma, Palmoplantar; Epidermolysis Bullosa; Ectodermal Dysplasia; Basal Cell Nevus Syndrome; Birt-Hogg-Dube Syndrome; Tuberous Sclerosis; Xeroderma Pigmentosum; Cutis Laxa; Albinism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Keratinisation disorders: Keratinisation disorders comprise a heterogeneous group characterised by abnormal epidermal differentiation, such as variants of ichthyosis and palmoplantar keratoderma.
- Skin fragility disorders: Skin fragility disorders comprise a group of inherited blistering diseases, such as variants of epidermolysis bullosa.
- Ectodermal dysplasias: Ectodermal dysplasias consists of multiple inherited disorders that are characterised by abnormalities of the embryonic ectoderm, such as hair, nails, sweat glands or teeth.
- Dermato-oncogenetic syndromes: This group are genodermatoses associated with the development of malignancies ((non-)cutaneous), such as basal cell nevus syndrome (BCNS), Birt-Hoog-Dubé syndrome, tuberous sclerosis, etc.
- Other genodermatoses: In this group genodermatoses are listed that do not fit the other groups as mentioned above, for example albinism and cutis laxa.

SUMMARY:
The goal of this observational study is to learn about the indications for prenatal diagnostics and preimplantation genetic testing for patients/couples affected by an inherited skin disease, and evaluate the clinical outcomes of these reproductive options. By providing a complete overview, the investigators aim to improve reproductive counselling for these patients/couples with a desire to have children.

To achieve this, the investigators aim to retrospectively collect data from a cohort of patiens/couples affected by an inherited skin disease on a national level (in the Netherlands) and also an international level from various countries in Europe.

ELIGIBILITY:
Inclusion Criteria:

* Couples affected with molecularly confirmed genodermatosis (i.e., keratinisation disorders, skin fragility diseases, ectodermal dysplasias, dermato-oncological syndromes, other genodermatoses)
* Prenatal diagnosis (PND) was performed and/or in vitro fertilisation (IVF) with pre-implantation genetic testing was performed (PGT).

Exclusion Criteria:

* No exclusion criteria were formulated.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of couples or adult inidividuals with genodermatosis keratinisation disorders, skin fragility diseases, ectodermal dysplasias, dermato-oncological syndromes, other genodermatoses) and a desire to have children, where PND and/or PGT were considered and/or performed.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of clinical outcomes of reproductive options | 2-3 years
  Outcomes of reproductive options such as prenatal diagnostics (PND) and preimplantation genetic testing (PGT) will be assessed, looking at indications, decision-making by professionals and/or the Dutch national indication committee as to whether or not to start a PGT procedure. The results of PND and PGT, pregnancy outcomes (success rates) and risks (i.e. the risk of miscarriage) will be summarised. The percentage of continuing pregnancies from prenatal screening techniques (especially PGT) will be calculated. In addition, the percentage of affected embryos will be calculated for different genodermatoses per PGT cycle using using the following formula: (number of affected embryos)/(total number of embryos)*100%.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Gostynski, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands